CLINICAL TRIAL: NCT07009678
Title: LOwer vs Upper Extremity Injection Agitated Saline for identifiCation of pATent Foramen ovalE (LOCATE) Pilot Study to Determine Safety of Lower Extremity Injection of Agitated Saline for Echocardiography of the Heart
Brief Title: Comparison of Lower vs Upper Extremity Injection Agitated Saline to Identify Patent Foramen Ovale With Echocardiography
Acronym: LOCATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. John's Hospital (Other)
Collaborators: University of Minnesota (Other); W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LOCATE Study 2023
Record Dates: First submitted 2025-05-12; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Patent Foramen Ovale; Cryptogenic Stroke; Embolic Infarction
MeSH Terms: conditions — Foramen Ovale, Patent; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Lower extremity used for injection of agitated saline to detect PFO (Experimental)
  Interventions: Diagnostic Test: intravenous access in greater saphenous vein compared to upper extremity site.

INTERVENTIONS:
Diagnostic Test: intravenous access in greater saphenous vein compared to upper extremity site. — Ultrasound access of greater saphenous vein with placement of midline 4French catheter and use of sphygmomanometer to regulate valsalva maneuver, imaging with and without valsalva and injection of agitated saline.
  Other Names: agitated saline injection (bubble study)

SUMMARY:
Study Title LOwer vs upper extremity injection agitated saline for identifiCation of pATent foramen ovalE (LOCATE) Pilot study to determine safety of lower extremity injection of agitated saline for echocardiography of the heart.

Primary Investigator Carmelo Panetta, MD University of Minnesota Physicians, St. John's Hospital 1600 St. Johns Blvd, suite 200, Maplewood, MN 55109

Study Design Prospective study of the safety and efficacy upper versus lower extremity injection agitated saline (bubble study) to identify patent foramen ovale (PFO) with echocardiography

Study Objective PFO are not identified in up to one quarter of subjects who have upper arm injection compared to femoral vein injection. We propose use of the PICC line nurses to obtain access in the greater saphenous vein in the lower leg and compare to the upper extremity injection in those subjects with concern for paradoxical embolus but previously PFO was not identified with an upper arm injection.

Study Endpoint Study the safety and efficacy of lower versus upper extremity injection agitated saline (bubble study) for identifying PFO

Subject Population Subjects with history of cryptogenic stroke or arterial embolus of unknown source with negative upper extremity injection agitate saline (bubble study) to identify a PFO.

Number of Sites Three sites to enroll subjects: St. John's/Woodwinds Hospital, University of Minnesota Medical Center and Southdale Hospital. One site to perform procedure at St John's hospital

Expected Time to Complete Enrollment 8-12 months

Schedule of Events Screening and consent of subjects who with negative bubble study for PFO to have upper and lower extremity bubble study, one week follow up and review echocardiography by two cardiologists.

Additional Information Data safety monitoring board will oversee the results every quarter Sample size 20 subjects were consented and enrolled is supported by this grant from GORE Medical.

DETAILED DESCRIPTION:
1. Introduction 1.1. Patent foramen ovale (PFO) is present in one third of the population based on autopsy (1) and up to half of those with a prior stroke (2). Diagnosis with echocardiography with an injection of agitated saline (bubble study) in the upper arm for detecting a PFO is the standard of care (3,4).

   1.2. Historical Treatments The presence of eustachian ridge in the right atrium is thought to direct blood flow from inferior vena cava (IVC) across the PFO. Conversely, the superior vena cava (SVC) has blood flow directed into the right ventricle. Three studies found in the cardiac catheterization laboratory the femoral vein injection agitated saline can identify up to one quarter more PFO than upper extremity injection(5-7). A larger recent study on 244 people already diagnosed with a PFO, found operators did not detect 25% of patients with PFO by upper arm injection agitated saline compared to femoral vein injection (7). A prospective multicenter study to compare upper arm versus the greater saphenous vein of the leg injection agitated saline with echocardiography to screen for PFO in subjects with prior cryptogenic stroke and of whom no PFO was detected via standard approach with the upper arm injection agitated saline. Funding available enroll 20 subjects with support from GORE therapeutics.

   1.3. Study Device Description Access in the greater saphenous vein for an agitated saline injection to identify more PFO compared to an upper arm injection.
2. Study Objectives 2.1. Primary Objective: 2.1.1. To evaluate the safety of access in the greater saphenous vein 2.1.2. To compare the efficacy and grading of size of a PFO from upper and lower extremity injection of agitated saline (bubble study
3. Study Design

3.1. Coordinators/leadership team: Primary Investigator: Carmelo Panetta, MD Admin lead for Clinical Research East Campus: Andrew Snyder Admin lead for Clinical Research UofMN Campus: Michelle Hintz Admin lead for Nursing team for central iv access/PICC line: Melissa Bustamonte Biostatistician: Sue Duval, PhD Professor of Medicine, Cardiovascular Division, UofMN

Fairview East Campus St. John's Hospital 1575 Beam Ave, Maplewood, MN 55109 Site Primary Investigator: Carmelo Panetta, MD, Adjunct Assistant Professor of Medicine, Cardiovascular Division, UofMN Non invasive/Echocardiography Director: Mitch Timmons, MD

University of Minnesota Medical Center 500 SE Harvard St, Minneapolis, MN 55455 Site Primary Investigator: Ganesh Raveendran, MD Professor of Medicine, Cardiovascular Division, UofMN Non invasive Director: Marc Pritzker, MD, Professor of Medicine, Cardiovascular Division, UofMN

Southdale Medical Center 6401 France Ave South, Edina, MN 55435 Site Primary Investigator: Marit Thorsgard, MD, Cardiology University of Minnesota Physicians

3.2. Description of Study Design This a prospective non-randomized multicenter study comparing upper versus lower extremity injection of agitated saline (bubble study) to identify PFO.

Subjects with history of cryptogenic stroke are screened who have negative bubble study for PFO by clinical research staff. Subjects are contacted and consented. Patients enrolled would be scheduled in the set times (currently allotted time slot in the afternoon Monday thru Friday at St.John's Hospital).

Access of the femoral vein is considered a procedure limited to the cardiac catheterization laboratory, intensive care unit or the emergency department and generally performed by a physician. The greater saphenous vein courses along the medial aspect of the thigh and enters the femoral vein near the femoral head (see Figure). The location of the greater saphenous vein is ideal for peripheral access given fewer valves to obstruct passage of bubbles to the heart, located usually 0.5 to 2 cm under the skin and is not associated with an artery. The nurse who is previously trained as a specialist in central intravenous access (often referred to as the peripherally inserted central catheter (PICC) line nurse) would be trained on locating and inserting a 4F (1.33mm diameter) 20cm length catheter (Bard MidLine catheter kit) into the greater saphenous vein in the thigh with standard sterile technique and ultrasound. The upper extremity peripheral intravenous line would be placed by echo technician or PICC nurse per standard of care.

After proper echocardiographic windows have been located, an injection of agitated saline and echocardiography would be performed to search for evidence of bubbles traversing from the right to the left atria and identifying a PFO. The identical agitated saline injection would then be done in lower extremity (which is then lifted up to help with flow back to the heart). After each injection, a waiting period to allow bubbles to pass thru the pulmonary circuit before the next injection. Standard views would be performed in each case to allow echocardiography reviewers to properly comment on the presence or absence of PFO.

The sheath/catheter in greater saphenous vein would be removed and manual pressure held to prevent bleeding for 15 minutes in the cardiac catheterization laboratory recovery suite.

Interpretation by two cardiologists would be completed (*one at the institution where the procedure performed and second outside cardiologist). The results would be placed into the electronic medical records and forwarded to the original physician who ordered the initial bubble study prior to enrollment in the LOCATE study.

ELIGIBILITY:
4.2. Inclusion Criteria

The subject is / has:

1. Age ≥18 at the time of informed consent signature.
2. Capable of complying with protocol requirements, including follow-up.
3. A Consent Form signed by Subject or legal representative.
4. Subjects have a history of concern for right to left shunt, such as a paradoxical embolus as source of a cryptogenic CVA requiring transthoracic echocardiography with agitated saline injection (bubble study)
5. No evidence of right to left shunt on injection of upper extremity using transthoracic echocardiography within the previous 24 months
6. If taking warfarin, patient is eligible if clinically able to hold warfarin for 3 days prior to procedure.

4.3. Exclusion Criteria

The subject is / has:

1. Enrolled in another drug or medical device study within 30 days of study enrollment.
2. Absence or size < 2mm diameter of both greater saphenous veins
3. Depth of the greater saphenous vein is > 3cm from the skin surface
4. Presence of deep vein thrombosis in either greater saphenous veins
5. Platelet count less than 50,000
6. International Normalized Ratio (INR) > 3 or liver failure within the last 6 months,
7. Taking oral anticoagulant (DOAC) within 24 hours
8. Taking high dose anticoagulation with heparin or low molecular weight heparin within 12 hours
9. Absence of adequate windows for echocardiographic imaging to detect shunt
10. Subject is unable to sign consent or considered a part of a vulnerable population: children/minors or age < 18 years, pregnant women, prisoners, terminally ill, comatose, intellectually challenged individuals who are assigned a guardian, institutionalized individuals, visual or hearing impaired without therapy to overcome the impairment, refugees.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy of placement of access in greater saphenous vein and performing agitated saline injection (bubble study) with echocardiography to screen for patent foramen ovale. | total time for procedure is 4 hours from arrival to departure. Follow up one week later to identify complications
  Placement of midline PICC line 4French in greater saphenous vein by PICC nurses with ultrasound and 18 gauge iv in right arm
Comparison of injection of agitate saline via upper versus lower extremity for detection of patent foramen ovale with echocardiography | A total time of two hours for the procedure and additional 30 minutes to call the participant one week after the procedure.
  see published manuscript - technique noted above.

SECONDARY OUTCOMES:
Injection of agitated saline via greater saphenous vein compared to upper arm injection for visualization of PFO | Two hours to do the echocardiography and additional 30 min to call the participant one week after the procedure.
  view the atria, septum and ventricles via three views with echocardiography. see published manuscript for details

CONTACTS AND LOCATIONS:
Locations (1):
- St. John's hospital, Maple Grove, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Panetta CJ, Forgosh LB, Bisinov E, Hussein H, Benditt D, Miller B, Yanavitski M, Thorsgard M, Jorgenson B, Raveendran G, Iqbal N. Lower vs upper extremity injection of agitated saline for identification of patent foramen ovale (LOCATE). J Echocardiogr. 2025 Sep;23(3):188-195. doi: 10.1007/s12574-025-00685-z. Epub 2025 Mar 22. PMID 40120067
- See also: Related Info — https://link.springer.com/article/10.1007/s12574-025-00685-z